CLINICAL TRIAL: NCT03978715
Title: The Effect of Implementing a Limb Loss Prevention Program on Amputation Rates
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Other Study IDs: 2018-0158
Record Dates: First submitted 2019-05-17; First posted 2019-06-07 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention-retrospective study — This is a retrospective study. No intervention
  Other Names: Retrospective study

SUMMARY:
The investigators plan to do a retrospective chart review on patients admitted to Parkland Hospital with diabetic foot infections, ulcers, and bone injuries from 2005 (5 years prior to the start of the diabetic limb preservation team) to present day. The investigators will collect information on demographics, medical/surgical history, social history, medications, laboratory results, peripheral arterial disease, wound severity, and treatment factors such as type of antibiotics, off-loading, debridement, wound healing, surgery interventions, complications, recurrence, and history and physical characteristics and exam from inpatient and outpatient encounters. This will be identified by current procedural terminology (CPT) codes for foot and leg amputations, and lower extremity revascularization procedures. Clinic visits will be identified to podiatry/foot wound, vascular surgery, invasive cardiology, general surgery, and physical therapy wound care in addition to inpatient encounters of these patients to determine the full scope of care received and to compare resources utilization before and after implementation of the diabetic limb preservation team.

DETAILED DESCRIPTION:
This will be a retrospective chart review on patients admitted to Parkland Hospital with diabetic foot infections, ulcers, and bone injuries from 2005 (5 years prior to the start of the diabetic limb preservation team) to present day. The investigators will collect information from medical records on demographics, medical/surgical history, social history, medications, laboratory results, peripheral arterial disease, wound severity, and treatment factors such as type of antibiotics, off-loading, debridement, wound healing, surgery interventions, complications, recurrence, and history and physical characteristics and exam from inpatient and outpatient encounters. This will be identified by current procedural terminology (CPT) codes for foot and leg amputations, and lower extremity revascularization procedures. Clinic visits will be identified to podiatry/foot wound, vascular surgery, invasive cardiology, general surgery, and physical therapy wound care in addition to inpatient encounters of these patients to determine the full scope of care received and to compare resources utilization before and after implementation of the diabetic limb preservation team. Study records will by a study identification number that will be assigned to the subject as soon as data collection is completed on each individual chart.

Non-parametric statistical analyses comparing individuals within each group and also differences between the groups will be performed using IBM SPSS Statistics version 25 (IBM Corporation, Armonk, New York).

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to Parkland Hospital with diabetic foot infections, ulcers, and bone injuries from 2005 (5 years prior to the start of the diabetic limb preservation team) to present day.

Exclusion Criteria:

* not fitting inclusion criteria.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to Parkland Hospital with diabetic foot infections, ulcers, and bone injuries from 2005 (5 years prior to the start of the diabetic limb preservation team) to present day.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
number of lower limb complications | One year
  The number of lower limb complications per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. in 2012. Diabetes Care. 2013 Apr;36(4):1033-46. doi: 10.2337/dc12-2625. Epub 2013 Mar 6. PMID 23468086
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. In 2007. Diabetes Care. 2008 Mar;31(3):596-615. doi: 10.2337/dc08-9017. PMID 18308683
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] Prompers L, Huijberts M, Apelqvist J, Jude E, Piaggesi A, Bakker K, Edmonds M, Holstein P, Jirkovska A, Mauricio D, Ragnarson Tennvall G, Reike H, Spraul M, Uccioli L, Urbancic V, Van Acker K, van Baal J, van Merode F, Schaper N. High prevalence of ischaemia, infection and serious comorbidity in patients with diabetic foot disease in Europe. Baseline results from the Eurodiale study. Diabetologia. 2007 Jan;50(1):18-25. doi: 10.1007/s00125-006-0491-1. Epub 2006 Nov 9. PMID 17093942
- [Background] Lavery LA, Peters EJ, Armstrong DG, Wendel CS, Murdoch DP, Lipsky BA. Risk factors for developing osteomyelitis in patients with diabetic foot wounds. Diabetes Res Clin Pract. 2009 Mar;83(3):347-52. doi: 10.1016/j.diabres.2008.11.030. Epub 2008 Dec 30. PMID 19117631
- [Background] Wukich DK, Hobizal KB, Sambenedetto TL, Kirby K, Rosario BL. Outcomes of Osteomyelitis in Patients Hospitalized With Diabetic Foot Infections. Foot Ankle Int. 2016 Dec;37(12):1285-1291. doi: 10.1177/1071100716664364. Epub 2016 Aug 22. PMID 27553085
- [Background] Mutluoglu M, Sivrioglu AK, Eroglu M, Uzun G, Turhan V, Ay H, Lipsky BA. The implications of the presence of osteomyelitis on outcomes of infected diabetic foot wounds. Scand J Infect Dis. 2013 Jul;45(7):497-503. doi: 10.3109/00365548.2013.765589. Epub 2013 Feb 5. PMID 23384323
- [Background] Lavery LA, Armstrong DG, Wunderlich RP, Tredwell J, Boulton AJ. Diabetic foot syndrome: evaluating the prevalence and incidence of foot pathology in Mexican Americans and non-Hispanic whites from a diabetes disease management cohort. Diabetes Care. 2003 May;26(5):1435-8. doi: 10.2337/diacare.26.5.1435. PMID 12716801
- [Background] Lavery LA, Lavery DC, Hunt NA, La Fontaine J, Ndip A, Boulton AJ. Amputations and foot-related hospitalisations disproportionately affect dialysis patients. Int Wound J. 2015 Oct;12(5):523-6. doi: 10.1111/iwj.12146. Epub 2013 Sep 19. PMID 24103293